CLINICAL TRIAL: NCT01505946
Title: Thrombin Generation Assay (TGA) as Predictive Test for Haemostatic Effectiveness of Factor VIII (FVIII) Concentrates in Patients Affected by Inherited Haemophilia A With FVIII Inhibitors High and Low Anamnestic Response.
Brief Title: Thrombin Generation Assay (TGA) as Predictive Test for Haemostatic. Effectiveness of FVIII Concentrates in Haemophiliac A With Inhibitors
Acronym: PredicTGA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Grifols Italia S.p.A (Industry)
Collaborators: Thrombinoscope (Unknown)
Responsible Party: Sponsor
Other Study IDs: PredicTGA; 373 (Other: Italian RSO http://osservazionali.agenziafarmaco.it)
Record Dates: First submitted 2012-01-05; First posted 2012-01-09 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Severe Hemophilia A With Inhibitor
Keywords: Thrombin; Hemophilia; Inhibitors; Immunotolerance; Haemostatic; FVIII; Epitopes; Moderately severe Hemophilia A with inhibitor
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- LOW RESPONDERS: Documented low anamnestic response after FVIII exposure (FVIII inhibitors titre >0.6 and < 5 BU/ml tested by Bethesda assay, Nijmegen modification). Patients who have never been submitted to ITI and also those patients who have completed ITI with partial success (defined as inhibitors titre >0.6 and < 5 BU/ml and no increase in the INH titer > 5 BU over treatment with FVIII)
  Interventions: Other: TGA (Thrombin generation Assay)
- HIGH RESPONDERS: Patients who documented high response after FVIII exposure (FVIII inhibitors titre > 5 BU/ml tested by Bethesda assay, Nijmegen modification) and who are potential candidates to a first or rescue ITI
  Interventions: Other: TGA (Thrombin generation Assay)

INTERVENTIONS:
Other: TGA (Thrombin generation Assay) — TGA will be performed on plasma in order to evaluate differences in the ability to stimulate the thrombin generation among the different class of FVIII concentrates and possibly identify the "most effective". The TGA will be quarterly repeated in order to verify if it is also adequate to check the therapy effectiveness during the study period

SUMMARY:
This is an observational, prospective, longitudinal, multicenter, cohort study designed with the scope to verify whether or not TGA may predict effectiveness of different FVIII concentrates class (devoid or rich of VWF) in patient affected by severe or moderately severe inherited haemophilia A and inhibitors.

DETAILED DESCRIPTION:
Rationale:

Hemophilia A is a serious and common hereditary bleeding disorder caused by deficiency of coagulation factor VIII (FVIII). Patients with this disease are treated with recombinant factor VIII or factor VIII concentrates derived from plasma.

Administration of exogenous FVIII in 15-35% of cases, cause the formation of antibodies to FVIII (inhibitors) that neutralize the activity of factor VIII, making the treatment ineffective.The development of inhibitors of factor VIII (FVIII) is the most serious and challenging complication of the treatment of hemophilia A and represents the highest economic burden for a chronic disease. Therefore, research is making great efforts to optimize the best therapeutic approach for the disease.

It has been observed that FVIII inhibitors display a wide range of immunoreactivity when tested against different classes of FVIII concentrates (with/without von Willebrand factor -VWF). It has been demonstrated that the different inhibitors reactivity may correlate with different ability of inhibitors to impair thrombin generation, as tested by Thrombin Generation Assay (TGA). In these patients TGA assay might be a tool to predict which FVIII concentrate has the greater haemostatic effectiveness.

It is also uncertain if the different classes of FVIII used in ITI protocols may have a different effectiveness in reducing the occurrence of BT bleedings and if this may correlate to lower reactivity, epitope specificity, VWF content and may be predicted by TGA. It would be very helpful to be able to give an evidence based diagnostic and prognostic instrument, the TGA, to aid physician to optimize the therapy for all inhibitors patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of inherited, severe (FVIII:C < 1%) or moderately severe haemophilia A (FVIII ≤ 2%)
* Any age
* Ability to comply with study methods and willingness to participate to the study
* Written informed consent.

FOR THE LOW RESPONDERS COHORT

- Documented low anamnestic response after FVIII exposure (FVIII inhibitors titre >0.6 and < 5 BU/ml tested by Bethesda assay, Nijmegen modification). It will be included in this study those patients who have never been submitted to ITI and also those patients who have completed ITI with partial success (defined as inhibitors titre >0.6 and < 5 BU/ml and no increase in the INH titer > 5 BU over treatment with FVIII)

INCLUSION CRITERIA FOR THE HIGH RESPONDERS COHORT

* Documented high response after FVIII exposure (FVIII inhibitors titre > 5 BU/ml tested by Bethesda assay, Nijmegen modification). It will be included in this study those patients who are potential candidates to a first or rescue ITI.
* Any historical peak ≥ 5 BU

Exclusion Criteria:

* Diagnosis of acquired haemophilia
* Diagnosis of inherited mild haemophilia A (FVIII > 2%)
* Life expectancy lower than 1 year
* Psychiatric illness and any other conditions may impair ability to comply with study methods

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with moderate or severe hemophilia A with inhibitors divided into two groups:
  1. Patients with inhibitors to FVIII and low anamnestic response: Low responders cohort
  2. Patients with inhibitors to FVIII and high anamnestic response: High responders cohort
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2012-03; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Thrombin generation result | 12 months
  Thrombin generation results of the TGA applied on plasma patients whith inhibitor matched with different class of FVIII concentrate

SECONDARY OUTCOMES:
Epitope mapping results | 12 months
  epitope mapping test on the plasma patient during the therapy for a follow-up period of 12 month
Incidence of all breakthrough (BT) bleedings | 12 months
  events/month
Total FVIII dose required to treat the patients | 12 months
  (IU/year)
the inhibitor titre course | 12 months
Use of bypassing agents | 12 months
  incidence of BT bleedings who require bypassing agents (events/months) average dose of bypassing agents (or days of treatment) needed to treat BT bleedings total dose of bypassing agent (and days of treatment) required overall (IU/year) and (days of treatment/year)
ITI outcome only for patient under this kind of treatment | 3 years
  % of Success (total, partial success or failure will be defined as in ITI study protocol) Time to tolerance (months), defined as the time to ITI success (total/partial)

CONTACTS AND LOCATIONS:
Overall Officials: Elena Santagostino, MD, PhD, Principal Investigator — Angelo Bianchi Bonomi" Haemophilia Thrombosis Centre I.R.C.S.S. Maggiore Hospital and University of Milan Via Pace 9, 20122 Milan - Italy
Locations (15):
- Italy (15):
  - Azienda Ospedaliero Universitaria Consorziale Policlinico di Bari, Bari, Apulia
  - Ospedale Civile dell' Annunziata, Cosenza, Calabria
  - Az. Universitaria Policlinico "Federico II" Dip. Assist. di Clinica Medica, Napoli, Campania
  - UO Angiologia e Malattie della Coagulazione "Marino Golinelli" Az Osp. Policlinico S. Orsola Malpighi, Bologna, Emilia-Romagna
  - Azienda Ospedaliera "Santa Maria della Misericordia", Udine, Friuli Venezia Giulia
  - Ematologia Dipartimento di Biotecnologie Cellulari Università La Sapienza - Policlinico Umberto I, Rome, Lazio
  - Ospedale Pediatrico Bambino Gesù di Roma, Rome, Lazio
  - Università Cattolica - Policlinico A. Gemelli, Rome, Lazio
  - Centro di Riferimento Emostasi e Trombosi in età pediatrica Ospedale dei bambini G. Di Cristina, Palermo, Palermo
  - Azienda Ospedialiera Ospedale Infantile Regina Margherita - S.Anna, Turin, Piedmont
  - Ospedale Le Molinette "S. G. Battista", Turin, Piedmont
  - Agenzia per l'Emofilia Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
  - Az. Ospedaliera di Padova, Clinica Medica IIa, Padua, Veneto
  - Azienda Ospedaliera Univesitaria Integrata di Verona - Borgo Roma, Verona, Veneto
  - Dipartimento di Terapie Cellulari ed Ematologia Ospedale San Bortolo, Vicenza, Veneto

REFERENCES:
- [Background] Wight J, Paisley S. The epidemiology of inhibitors in haemophilia A: a systematic review. Haemophilia. 2003 Jul;9(4):418-35. doi: 10.1046/j.1365-2516.2003.00780.x. PMID 12828678
- [Background] Salvagno GL, Astermark J, Ekman M, Franchini M, Guidi GC, Lippi G, Poli G, Berntorp E. Impact of different inhibitor reactivities with commercial factor VIII concentrates on thrombin generation. Haemophilia. 2007 Jan;13(1):51-6. doi: 10.1111/j.1365-2516.2006.01400.x. PMID 17212725
- [Background] Iorio A, Halimeh S, Holzhauer S, Goldenberg N, Marchesini E, Marcucci M, Young G, Bidlingmaier C, Brandao LR, Ettingshausen CE, Gringeri A, Kenet G, Knofler R, Kreuz W, Kurnik K, Manner D, Santagostino E, Mannucci PM, Nowak-Gottl U. Rate of inhibitor development in previously untreated hemophilia A patients treated with plasma-derived or recombinant factor VIII concentrates: a systematic review. J Thromb Haemost. 2010 Jun;8(6):1256-65. doi: 10.1111/j.1538-7836.2010.03823.x. Epub 2010 Mar 17. PMID 20345722
- [Background] Astermark J, Santagostino E, Keith Hoots W. Clinical issues in inhibitors. Haemophilia. 2010 Jul;16 Suppl 5:54-60. doi: 10.1111/j.1365-2516.2010.02294.x. PMID 20590857
- [Background] Gringeri A, Mantovani LG, Scalone L, Mannucci PM; COCIS Study Group. Cost of care and quality of life for patients with hemophilia complicated by inhibitors: the COCIS Study Group. Blood. 2003 Oct 1;102(7):2358-63. doi: 10.1182/blood-2003-03-0941. Epub 2003 Jun 19. PMID 12816859
- [Background] Kopecky EM, Greinstetter S, Pabinger I, Buchacher A, Romisch J, Jungbauer A. Mapping of FVIII inhibitor epitopes using cellulose-bound synthetic peptide arrays. J Immunol Methods. 2006 Jan 20;308(1-2):90-100. doi: 10.1016/j.jim.2005.10.016. Epub 2005 Dec 5. PMID 16376372
- [Background] Chambost H. Assessing risk factors: prevention of inhibitors in haemophilia. Haemophilia. 2010 Mar;16 Suppl 2:10-5. doi: 10.1111/j.1365-2516.2009.02197.x. PMID 20132333
- [Background] Boekhorst J, Lari GR, D'Oiron R, Costa JM, Novakova IR, Ala FA, Lavergne JM, VAN Heerde WL. Factor VIII genotype and inhibitor development in patients with haemophilia A: highest risk in patients with splice site mutations. Haemophilia. 2008 Jul;14(4):729-35. doi: 10.1111/j.1365-2516.2008.01694.x. Epub 2008 May 12. PMID 18503540
- [Background] Coppola A, Margaglione M, Santagostino E, Rocino A, Grandone E, Mannucci PM, Di Minno G; AICE PROFIT Study Group. Factor VIII gene (F8) mutations as predictors of outcome in immune tolerance induction of hemophilia A patients with high-responding inhibitors. J Thromb Haemost. 2009 Nov;7(11):1809-15. doi: 10.1111/j.1538-7836.2009.03615.x. Epub 2009 Sep 9. PMID 19740093
- [Background] Kallas A, Talpsep T. von Willebrand factor in factor VIII concentrates protects against neutralization by factor VIII antibodies of haemophilia A patients. Haemophilia. 2001 Jul;7(4):375-80. doi: 10.1046/j.1365-2516.2001.00530.x. PMID 11442642
- [Background] Astermark J, Voorberg J, Lenk H, DiMichele D, Shapiro A, Tjonnfjord G, Berntorp E. Impact of inhibitor epitope profile on the neutralizing effect against plasma-derived and recombinant factor VIII concentrates in vitro. Haemophilia. 2003 Sep;9(5):567-72. doi: 10.1046/j.1365-2516.2003.00802.x. PMID 14511295
- [Background] Berntorp E. Variation in factor VIII inhibitor reactivity with different commercial factor VIII preparations: is it of clinical importance? Haematologica. 2003 Jun;88(6):EREP03. PMID 12826529
- [Background] Gringeri A. VWF/FVIII concentrates in high-risk immunotolerance: the RESIST study. Haemophilia. 2007 Dec;13 Suppl 5:73-7. doi: 10.1111/j.1365-2516.2007.01579.x. PMID 18078402
- [Background] Goudemand J, Rothschild C, Demiguel V, Vinciguerrat C, Lambert T, Chambost H, Borel-Derlon A, Claeyssens S, Laurian Y, Calvez T; FVIII-LFB and Recombinant FVIII study groups. Influence of the type of factor VIII concentrate on the incidence of factor VIII inhibitors in previously untreated patients with severe hemophilia A. Blood. 2006 Jan 1;107(1):46-51. doi: 10.1182/blood-2005-04-1371. Epub 2005 Sep 15. PMID 16166584
- [Background] Gringeri A, Monzini M, Tagariello G, Scaraggi FA, Mannucci PM; Emoclot15 Study Members. Occurrence of inhibitors in previously untreated or minimally treated patients with haemophilia A after exposure to a plasma-derived solvent-detergent factor VIII concentrate. Haemophilia. 2006 Mar;12(2):128-32. doi: 10.1111/j.1365-2516.2006.01201.x. PMID 16476086
- [Background] Kurth MA, Dimichele D, Sexauer C, Sanders JM, Torres M, Zappa SC, Ragni M, Leonard N. Immune tolerance therapy utilizing factor VIII/von Willebrand factor concentrate in haemophilia A patients with high titre factor VIII inhibitors. Haemophilia. 2008 Jan;14(1):50-5. doi: 10.1111/j.1365-2516.2007.01560.x. Epub 2007 Oct 18. PMID 17941829
- [Background] Orsini F, Rotschild C, Beurrier P, Faradji A, Goudemand J, Polack B. Immune tolerance induction with highly purified plasma-derived factor VIII containing von Willebrand factor in hemophilia A patients with high-responding inhibitors. Haematologica. 2005 Sep;90(9):1288-90. PMID 16154861
- [Background] Gringeri A, Musso R, Mazzucconi MG, Piseddu G, Schiavoni M, Pignoloni P, Mannucci PM; RITS-FITNHES Study Group. Immune tolerance induction with a high purity von Willebrand factor/VIII complex concentrate in haemophilia A patients with inhibitors at high risk of a poor response. Haemophilia. 2007 Jul;13(4):373-9. doi: 10.1111/j.1365-2516.2007.01484.x. PMID 17610550